CLINICAL TRIAL: NCT03418090
Title: Evaluation of Hyperpolarized 129Xe MRI as Compared to 133Xe Scintigraphy for the Assessment of Pulmonary Function in Patients Being Evaluated for Possible Lung Transplant Surgery
Brief Title: Hyperpolarized Xenon MRI for Assessment of Pulmonary Function in Lung Transplant
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Polarean, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: POL-Xe-002
Record Dates: First submitted 2018-01-25; First posted 2018-02-01 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Pulmonary Surgical Procedures

STUDY DESIGN:
Intervention Model Description: Open label crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Active Comparator): Subjects will first undergo hyperpolarized 129Xe MRI followed by 133Xe scintigraphy
  Interventions: Drug: 129Xe MRI; Drug: 133XE scintigraphy
- Arm 2 (Active Comparator): Subjects will first undergo 133Xe scintigraphy followed by hyperpolarized 129Xe MRI
  Interventions: Drug: 129Xe MRI; Drug: 133XE scintigraphy

INTERVENTIONS:
Drug: 129Xe MRI — Evaluation of pulmonary function
  Other Names: 129Xenon MRI
Drug: 133XE scintigraphy — Evaluation of pulmonary function
  Other Names: 133Xenon scintigraphy

SUMMARY:
This study compares the equivalence of hyperpolarized 129Xe MRI to 133Xe scintigraphy for the evaluation of pulmonary function in patients being evaluated for lung transplant.

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label, cross-over Phase 3 study evaluating hyperpolarized 129Xe gas MRI as compared to 133Xe scintigraphy for the evaluation of pulmonary function. This study will enroll subjects being evaluated for possible lung transplant surgery (either single or bilateral) . Subjects will have both a 129Xe MRI and 133Xe scintigraphy image. The vast differences in technique for obtaining hyperpolarized 129Xe MRI as compared to 133Xe scintigraphy make it impossible to blind study procedures. However, all image interpretation will be performed by personnel blinded to the subject's medical history and all study assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥18 years of age.
2. Subject is being evaluated for possible lung transplant surgery (either single or bilateral).
3. Subject is able to undergo MRI imaging and able to fit in the MRI coil.
4. Subject is willing and able to comply with all study procedures.
5. Subject must understand and voluntarily sign an informed consent form (ICF) prior to any study specific assessments or procedures.

Exclusion Criteria:

1. Baseline blood oxygen saturation (SpO2) <90% at rest. For subjects requiring routine supplemental oxygen, SpO2 measurements should be taken with the patient's normal oxygen supplementation.
2. Subjects that have undergone a prior pneumonectomy surgery to either lung.
3. Female subjects of childbearing potential with a positive serum pregnancy test at screening, or who are not taking (or not willing to take) acceptable birth control measures through the Follow-up Period. Adequate birth control methods include with a monogamous partner who was sterilized more than 6 months prior to screening, or measures with a Pearl index of <1 used consistently and correctly (including intrauterine devices, or implantable, injectable, oral, or transdermal contraceptives). Women are not considered to be of childbearing potential if they meet at least 1 of the following 2 criteria as documented by the Investigator:

   * They have had a hysterectomy, bilateral salpingectomy, or bilateral oophorectomy at a minimum of 1 menstrual cycle prior to signing the ICF; or
   * They are post-menopausal: for women ≥55 years of age, defined as ≥1 year since their last menstrual period, or for women <55 years of age, defined as ≥1 year since their last menstrual period and have a follicle-stimulating hormone (FSH) level in the laboratory's normal range for post-menopausal phase.
4. Women who are lactating and insist on breast feeding.
5. Have received any other investigational therapy within 4 weeks prior to Screening.
6. Requires anesthesia or heavy sedation to undergo MRI testing. Mild sedation could be acceptable (i.e. a low dose oral acting anxiolytic medication such as alprazolam) as long as, in the opinion of the investigator, the subject meets Inclusion Criteria #4 and #5.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
Right lung function | 48 hours
  Scan predicted contribution of right lung to overall lung function

SECONDARY OUTCOMES:
6 zone analysis | 48 hours
  The percentage function contributed by each of the individual 6 lung zones.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth P West, Study Director — Polarean, Inc.
Locations (2):
- United States (2):
  - Duke University Hospital, Durham, North Carolina
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Undecided